CLINICAL TRIAL: NCT06504485
Title: Immunological and Virological Characterization of Patients With Chronic HBV-HDV Infection: Association With Disease Outcomes and Response to Bulevirtide Treatment
Brief Title: Immunological and Virological Characterization of Patients With Chronic HBV-HDV Infection: Outcomes and Response to Bulevirtide Treatment
Acronym: MPR_BD
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: University of Milan (Other); Parma University Hospital (Other); University of Rome Tor Vergata (Other)
Responsible Party: Sponsor
Other Study IDs: P2022WEXP2
Record Dates: First submitted 2024-07-05; First posted 2024-07-16 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis D
MeSH Terms: conditions — Hepatitis D | interventions — bulevirtide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hepatis Delta naive: Patients with HDV infection naïve to Bulevirtide therapy
- Hepatis Delta in therapy: Patients with HDV cirrhosis consecutively started on Bulevirtide therapy during the study enrollment period
  Interventions: Drug: Bulevirtide

INTERVENTIONS:
Drug: Bulevirtide — dose of 2 mg/day subcutaneously
  Groups: Hepatis Delta in therapy

SUMMARY:
Pharmacological, single-center, non-profit observational study.

The present study is part of a cooperation project between the SC Gastroenterology and Hepatology, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico (Milan, Italy), the University of Milan, the University of Parma and Rome Tor Vergata, funded under the call for Research Projects of Significant National Interest - 2022 PNRR Call (Prot. P2022WEXP2).

Hepatitis D virus (HDV) is a defective RNA virus, which requires the presence of hepatitis B virus (HBV) to infect liver cells and propagate. To date, the mechanisms underlying the accelerated disease progression in the natural history of Delta hepatitis are poorly understood, as is the course of the HDV-specific immune response (CD4 and CD8 T cells). As in chronic HBV and HCV infections, the outcome of chronic HDV infection appears to be dictated primarily by the host immune response, which represents a key determinant for virus control or persistence. For HBV/HDV coinfection, the role of T cells has not been well defined, as suitable animal models are lacking and so far few HDV-specific T cell epitopes have been precisely mapped, mainly limited to HLA-B alleles.

The study is divided into two substudies (cross-sectional and longitudinal). The primary objective of the cross-sectional study is to calculate the prevalence of HDV-specific T responses in patients with chronic HBV-HDV infection naïve to treatment with Bulevirtide. The primary objective of the longitudinal study is the change in the prevalence of HDV-specific T responses in patients with chronic HBV-HDV infection during treatment with Bulevirtide compared to baseline (pre-treatment).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Ability to understand and sign the informed consent
* Chronic HDV infection defined by positivity of HBsAg antigen (HBV) and HDV RNA (HBV-HDV co-infection) for at least 6 months at the time of enrollment.

Exclusion Criteria:

* Co-infection with other viruses (HCV, HIV)
* Treatment with immunosuppressive/immunomodulatory drugs
* Other congenital and/or acquired immunodeficiency conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients co-infected with HBV-HDV (defined by positivity of HDV RNA for at least 6 months) who meet the inclusion criteria and no exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Calculate the prevalence of HDV-specific T responses in patients with chronic HBV-HDV infection naïve to treatment with Bulevirtide | through study completion, an average of 2 year
  Prevalence of HDV-specific T responses in patients with chronic HBV-HDV infection naïve to treatment with Bulevirtide
Change in the prevalence of HDV-specific T responses in patients with chronic HBV-HDV infection during treatment with Bulevirtide compared to baseline (pre-treatment) | Month 12
  Prevalence of HDV-specific T responses in patients with chronic HBV-HDV infection after 12 months of treatment with Bulevirtide compared to baseline (pre-therapy)

SECONDARY OUTCOMES:
Correlate HDV-specific T cell response with stage of liver disease | through study completion, an average of 2 year
  Correlation of HDV-specific T cell response with stage of liver disease
Analyze the role of new HBV serum biomarkers (HBcrAg, HBV RNA, HBsAg isoforms) in predicting the stage of liver disease | through study completion, an average of 2 year
  Quantification of new HBV serum biomarkers (HBcrAg, HBV RNA, HBsAg isoforms) and correlation with the stage of liver disease
Correlate the quantification of HDV RNA within exosomes with the stage of liver disease | through study completion, an average of 2 year
  Correlation between the quantification of HDV RNA within exosomes and the disease phenotype
Investigate the correlation between the genetic heritage of HDV and the stage of liver disease | through study completion, an average of 2 year
  Correlation between the genetic heritage of HDV and the stage of liver disease
Define the transcriptional and molecular signatures of CD8 T cell dysfunction in patients with chronic HBV/HDV coinfection | through study completion, an average of 2 year
  Transcriptional and molecular signatures of CD8 T cell dysfunction in patients with chronic HBV/HDV coinfection
Understanding the role of virus mutations in the virus's ability to escape CD8 T cell surveillance | through study completion, an average of 2 year
  Correlation between HDV mutations and the ability of the virus itself to escape CD8 T cell surveillance
Correlate the prevalence of HDV-specific T cell responses with response to treatment over time | Month 6
  Correlation between the change in HDV-specific T responses
Correlate the prevalence of HDV-specific T cell responses with response to treatment over time | Month 18
  Correlation between the change in HDV-specific T responses
Correlate the prevalence of HDV-specific T cell responses with response to treatment over time | through study completion, an average of 2 year
  Correlation between the change in HDV-specific T responses
Analyze the role of new HBV serum biomarkers (HBcrAg, HBV RNA, HBsAg isoforms) in predicting response to treatment with Bulevirtide; | through study completion, an average of 2 year
  Quantification of new HBV serum biomarkers (HBcrAg, HBV RNA, HBsAg isoforms) and correlation with response to treatment with Bulevirtide
Correlate quantification of HDV RNA within exosomes with response to Bulevirtide treatment | through study completion, an average of 2 year
  Correlation between the quantification of HDV RNA within exosomes and the response to treatment with Bulevirtide
Investigate the correlation between the genetic heritage of HDV and the response to treatment with Bulevirtide | through study completion, an average of 2 year
  Correlation between HDV genetic heritage and response to treatment with Bulevirtide

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation IRCCS Ca' Granda Ospedale Maggiore Policlinico, Division of Gastroenterology and Hepatology, Milan, Italy., Milan, Italy